CLINICAL TRIAL: NCT03773029
Title: Effects of Isoflavones on Cardiovascular Disease Risk Factors, Bone Metabolism Markers, Serum Concentrations of Fructoseamine and Advanced Glycated End Products in Peritoneal Dialysis Patients
Brief Title: The Effects of Isoflavones on Cardiovascular and Bone Metabolism Markers in Peritoneal Dialysis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Nutrition and Food Technology Institute (Other)
Responsible Party: Principal Investigator, zahra yari, Principal Investigator, National Nutrition and Food Technology Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1397.247
Record Dates: First submitted 2018-12-10; First posted 2018-12-12 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2018-12

CONDITIONS: Peritoneal Dialysis Patients
MeSH Terms: interventions — Soybean Proteins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- isoflavone (Active Comparator): 100 mg soy isoflavone (as 2 capsules)
  Interventions: Dietary Supplement: soy isoflavone
- control (Placebo Comparator): 2 capsules of placebo
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: soy isoflavone — 100 mg soy isoflavone (as 2 capsules)
  Arms: isoflavone
Other: placebo — 2 capsules of placebo
  Arms: control

SUMMARY:
The aim of this double-blind randomized clinical trial is to determine the effects of isoflavones on cardiovascular disease risk factors, bone metabolism markers, serum concentrations of fructoseamine and advanced glycated end products in peritoneal dialysis patients. Forty-four patients from shafa clinic and Dr.najafi's clinic will randomly assign to either isoflavone or placebo group. The patients in isoflavone group will receive 100 mg soy isoflavone (as 2 capsules) daily for 8 weeks, while the placebo group will receive identical placebo. At the baseline and the end of the study,7 ml blood will be collected from each patient after a 12-14-hours fasting and serum concentrations of Lp (a), MDA, hs-CRP, sICAM-1, bone alkaline phosphatase, osteocalcin, N-telopeptide, osteoprotegerin, RANKL, iPTH, triglyceride, total cholesterol, HDL-C, LDL-C, fructoseamine, carboxymethyl lysine, pentosidine, glucose, albumin, calcium and phosphorous will be measured. Furthermore, blood pressure measurements will be performed twice with a ten-minute interval between testing

ELIGIBILITY:
Inclusion Criteria:

Continuous Ambulatory Peritoneal Dialysis for 6 months or more Body mass index below 35

Exclusion Criteria:

infections inflammatory diseases; liver diseases; past medical history of cancer receiving glucocorticoid and anti-inflammatory drugs receiving isoflavone supplements Constant consumption of soy or foods containing soy in the diet

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Lp (a) | 8 weeks
  Serum concentrations of lipoprotein-a
MDA | 8 weeks
  Serum concentrations of malondialdehyde
hs-CRP | 8 weeks
  Serum concentrations of high sensitivity c-reactive protein
sICAM-1 | 8 weeks
  Serum concentrations of Soluble intercellular adhesion molecule-1
bone alkaline phosphatase | 8 weeks
  Serum concentrations of bone alkaline phosphatase
osteocalcin | 8 weeks
  Serum concentrations of osteocalcin
N-telopeptide | 8 weeks
  Serum concentrations of N-telopeptide
Osteoprotegerin | 8 weeks
  Serum concentrations of Osteoprotegerin
RANKL | 8 weeks
  Serum concentrations of Receptor activator of nuclear factor kappa-Β ligand
triglyceride | 8 weeks
  Serum concentrations of triglyceride
total cholesterol | 8 weeks
  Serum concentrations of total cholesterol
HDL-C | 8 weeks
  Serum concentrations of High-density lipoprotein cholesterol
LDL-C | 8 weeks
  Serum concentrations of low-density lipoprotein cholesterol
sVCAM-1 | 8 weeks
  Serum concentrations of Soluble vascular adhesion molecule-1
E-selectin | 8 weeks
  Serum concentrations of E-selectin

SECONDARY OUTCOMES:
albumin | 8 weeks
  Serum concentrations of albumin
calcium | 8 weeks
  Serum concentrations of calcium
phosphorous | 8 weeks
  Serum concentrations of phosphorous
iPTH | 8 weeks
  Serum concentrations of Intact parathyroid hormone

CONTACTS AND LOCATIONS:
Locations (1):
- National Nutrition and Food Technology Research Institute, Tehran, Iran (the Islamic Republic Of), Iran

REFERENCES:
- [Derived] Yari Z, Tabibi H, Najafi I, Hedayati M, Movahedian M. Effects of soy isoflavones on serum lipids and lipoprotein (a) in peritoneal dialysis patients. Nutr Metab Cardiovasc Dis. 2020 Jul 24;30(8):1382-1388. doi: 10.1016/j.numecd.2020.04.023. Epub 2020 May 5. PMID 32513581
- [Derived] Yari Z, Tabibi H, Najafi I, Hedayati M, Movahedian M. Effects of isoflavones on bone turnover markers in peritoneal dialysis patients: a randomized controlled trial. Int Urol Nephrol. 2020 Jul;52(7):1367-1376. doi: 10.1007/s11255-020-02523-w. Epub 2020 Jun 1. PMID 32488754